CLINICAL TRIAL: NCT04720027
Title: Long Term Outcomes of the Double Blind Randomised Controlled Trial of Radiofrequency Thermal Ablation Treatments of Great Saphenous Varicose Veins: Closurefast vs. RFITT vs. EVRF
Brief Title: Long Term Study of 3 Radiofrequency Devices
Acronym: 3RF-5Years
Status: Completed | Type: Observational
Sponsor: Worcestershire Acute Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: WorcestershireNHS
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Varicose Veins of Lower Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Closurefast: Patients who were randomised to and underwent radiofrequency ablation using the Closurefast device in the original 3RF Study
  Interventions: Diagnostic Test: Duplex imaging
- Radiofrequency Induced Thermal Therapy (RFITT): Patients who were randomised to and underwent radiofrequency ablation using the RFITT device in the original 3RF Study
  Interventions: Diagnostic Test: Duplex imaging
- EndoVenous Radiofrequency (EVRF): Patients who were randomised to and underwent radiofrequency ablation using the EVRF device in the original 3RF Study
  Interventions: Diagnostic Test: Duplex imaging

INTERVENTIONS:
Diagnostic Test: Duplex imaging — Completion of AVVQ and EQ5D questionnairs
  Other Names: Completion of Quality Of Life Questionnaires

SUMMARY:
To establish which of the radiofrequency venous ablation modalities studied in the original 3RF study (Venefit (Closurefast), vs. Radiofrequency induced Thermal Therapy vs. Endovenous Radiofrequency) is most effective in relieving patients' symptoms and signs from varicose veins disease, and in maintaining absence of reflux in the treated vein segment (of the great saphenous vein (GSV)) 5 years following surgery.

DETAILED DESCRIPTION:
Results of randomised trials and meta-analyses have shown that endovenous thermal ablation of the GSV using radiofrequency ablation or laser is associated with improved recovery compared with conventional surgery. Furthermore, radiofrequency ablation (using the Closurefast device) has been shown to cause less pain and require less analgesic intake than laser treatment. At the time the 3 RF study was conceived there were two other radiofrequency devices that were marketed to have theoretical advantages over the Closurefast technique. All three devices were in use in clinical practice (including at Worcestershire Royal Hospital) in 2013. The initial study focused on clinical results (up to 12 months) and anatomical results (up to 6 months) and remains the only clinical trial to date that has directly compared the outcomes of radiofrequency thermal ablation devices.

This second (long term) phase of the study aims to assess which of the radiofrequency venous ablation modalities studied in the original 3RF study (Venefit (Closurefast), vs. Radiofrequency induced Thermal Therapy vs. Endovenous Radiofrequency) is most effective in relieving patients' symptoms and signs from varicose veins disease, and in maintaining absence of reflux in the treated vein segment (of the great saphenous vein (GSV)) 5 years following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients originally recruited to and studied in the 3RF Study (clinicaltrials.gov identifier: NCT02441881) who give informed consent to take part in this long term study

Exclusion Criteria:

* Patients originally recruited to and studied in the 3RF Study (clinicaltrials.gov identifier: NCT02441881) who do not give informed consent to take part in this long term study

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The 180 patients who were originally recruited to and studied in the 3RF Study (clinicaltrials.gov identifier: NCT02441881)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Anatomical assessment of ablation of treated GSV segment | 5 years after treatment
  Aanatomical assessment of total ablation of treated segment will be assessed:
  Failure will be defined as any segment of the treated trunk (> 2cm from the saphenofemoral junction) that is patent (compressible) and demonstrates reflux (>1 second) on duplex scanning.

SECONDARY OUTCOMES:
Absence of recurrent varicose veins and or return of symptoms | 5 years after treatment
  Assessments using disease specific (AVVQ) and generic (EQ5D) quality of life scores by means of self-completed questionnaires completed at a single consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Nyamekye, FRCS, MD, Principal Investigator — Worcestershire Acute Hospitals NHS Trust
Locations (1):
- Worcestershire Acute Hospitals NHS Trust, Worcester, Worcestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not plan to share IPD

REFERENCES:
- [Background] Nyamekye IK, Dattani N, Hayes W, Harding D, Holloway S, Newman J. A Randomised Controlled Trial Comparing Three Different Radiofrequency Technologies: Short-Term Results of the 3-RF Trial. Eur J Vasc Endovasc Surg. 2019 Sep;58(3):401-408. doi: 10.1016/j.ejvs.2019.01.033. Epub 2019 Jul 24. PMID 31351832
- [Derived] Nyamekye IK, Pullen BJ, Kelly N, Hayes W. Six Year Extension Study of Patients From a Randomised Clinical Trial Comparing Venefit, Radiofrequency Induced Thermal Therapy, and Endovenous Radiofrequency Ablation for Treatment of Incompetent Great Saphenous Veins. Eur J Vasc Endovasc Surg. 2023 Jul;66(1):94-101. doi: 10.1016/j.ejvs.2023.03.021. Epub 2023 Mar 21. PMID 36958479